CLINICAL TRIAL: NCT06096467
Title: The Impact of Cross-disciplinary Teamwork Care Model and Exercise Intervention on Physical Function Falls, and Physical Restraint for Residents in Long-term Care Institution
Brief Title: The Impact of Exercise Intervention on Physical Function Falls, and Physical Restraint for Long-term Care Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardinal Tien Hospital (Other)
Responsible Party: Principal Investigator, Tsai Ren Jei, MS, Principal Investigator, Cardinal Tien Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: TSGHIRB SOP AF03-05.4/D6.0
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Exercise Intervention; Protein Supplementation
Keywords: protein supplementation; exercise; long-term care institutions
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehension exercise training combined with protein supplementation (CET+PS) (Experimental): CET+PS: the comprehension exercise training combined with protein supplementation
  Interventions: Behavioral: Comprehension Exercise Training; Dietary Supplement: Protein Supplement
- Comprehension exercise training combined with placebo milk (CET+PC) (Placebo Comparator): CET+PC: the comprehension exercise training combined with placebo milk
  Interventions: Behavioral: Comprehension Exercise Training; Dietary Supplement: Placebo milk

INTERVENTIONS:
Behavioral: Comprehension Exercise Training — Comprehension exercise: 45~50 minutes exercise for each session(warm-up, resistive, functional activities and balance exercise, and cool-down)
  Other Names: CET
Dietary Supplement: Placebo milk — Placebo milk: 8 g. protein for each serving and provided immediately after the CET session
  Other Names: PC
  Arms: Comprehension exercise training combined with placebo milk (CET+PC)
Dietary Supplement: Protein Supplement — Protein Supplement: 40 g. whey protein for each serving and provided immediately after the CET session
  Other Names: PS
  Arms: Comprehension exercise training combined with protein supplementation (CET+PS)

SUMMARY:
The goal of this clinical trial is to test the effect of the Cross-disciplinary Teamwork Care Model and Exercise Intervention in residents living in long-term care institutions. The main question[s] it aims to answer are:

* Increased physical performance.
* Reduced the physical restraint.
* Reduced fall accidents.

Participants will accept the comprehension Exercise Intervention combined with protein supplementation or not.

DETAILED DESCRIPTION:
The prevalence of institutional physical restraint, both at home and abroad, remains alarmingly high. The Health Care Financing Administration (HCFA) in 1999 provided a comprehensive definition for physical restraint in nursing homes, encompassing any manual, physical, or mechanically related device, material, or tool attached to or installed on a resident's body that hinders their freedom of movement or contact with their body. The primary objective of implementing physical restraint in healthcare settings is to prevent patients from becoming agitated, safeguard them from self-inflicted injuries, protect the staff, prevent falls, and manage routine care and behavior control. Unfortunately, falls are a common occurrence among the elderly, whether they are living at home or in institutional settings.

Falls in the elderly are often attributed to a myriad of factors, including poor physical function and the use of multiple medications. Impaired physical function components such as diminished muscle strength, imbalanced balance abilities, delayed reaction times, postural hypotension, and cognitive dysfunction are frequently observed contributors to falls. Furthermore, malnutrition or undernutrition is a prevalent concern among the elderly, affecting those being cared for at home or placed in institutional settings. Malnutrition compounds the adverse effects on physical function, leading to muscular weakness and potentially the development of sarcopenia, a condition characterized by a loss of muscle mass and strength. This not only compromises immunity but also elevates the risk of disease and increases the likelihood of disability or falls among the elderly.

In response to these challenges, this study aims to be conducted collaboratively by the three private nursing type centers (Guang-nenn Care Center for the Elderly, Tung-shin Long-term Care Center, and the Hu-An Long-term Care Center for the Elderly). The study will involve 22 elderly patients. The primary objective is to address the multifaceted issues of physical restraint, falls, and declining physical function in elderly care facilities.

The research team began by conducting a systematic review of the existing literature on long-term care institutions, interdisciplinary teamwork care models, sports interventions, physical function, falls, and physical restraint. This comprehensive review served as the foundation for designing a 12-month "comprehensive multi-component exercise" program. The program is based on evidence from the literature and aims to enhance the strength, balance, and mobility of residents through carefully tailored exercise interventions.

The ultimate goal of the exercise program is to reduce the utilization of physical restraint as a means to prevent falls. By focusing on improving residents' physical abilities, the research anticipates a decrease in the need for physical restraint, ultimately enhancing the quality of life for elderly individuals in these long-term care facilities.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 65 years or older
2. Placement is greater than or equal to 6 months
3. Less dependency in activities of daily life (ADL) function50 (severe to moderate dependency, Barthel index: 21 ≤ score ≤ 90)
4. Able to understand the exercise instructions and follow the order.

Exclusion Criteria:

1. Skeletomuscular (severe osteoarthritis (OA) or recent or mal- or non-union fracture, etc.) or cardiopulmonary diseases (COVID-19 or unstable angina or controlled hypertension, etc.) that are unstable and pose a threat to safety
2. Mental disorders that prevent the subject from following instructions (severe mental disorder, Short Portable Mental State Questionnaire (SPMSQ): 8 ≤ score ≤ 10).
3. Protein supplementations are contraindicated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | T1: before Phase 1 intervention; T2: immediately after Phase 1 intervention; T3: before Phase 2 intervention; T2: immediately after Phase 2 intervention, and completed the assessments within 1 week.
  To evaluate the physical functional performance of elderly individuals.The assessment primarily comprises three components: standing balance, mobility (four-meter walk test), and muscle strength (five-repetition sit-to-stand test).

SECONDARY OUTCOMES:
Muscle strength of Upper limb and lower limb | T1: before Phase 1 intervention; T2: immediately after Phase 1 intervention; T3: before Phase 2 intervention; T4: immediately after Phase 2 intervention, and completed the assessments within 1 week.
  Test the strength of hand grip and knee extension.
Functional forward reach (FFR) | T1: before Phase 1 intervention; T2: immediately after Phase 1 intervention; T3: before Phase 2 intervention; T4: immediately after Phase 2 intervention, and completed the assessments within 1 week.
  The Functional Forward Reach Test is used to assess subjects' standing balance.
Number of fall occurrences | T1: before Phase 1 intervention; T2: immediately after Phase 1 intervention; T3: before Phase 2 intervention; T4: immediately after Phase 2 intervention, and completed the assessments within 1 week.
  Read records from nursing care daily record the institutions.
Number of physical restraint occurrence | T1: before Phase 1 intervention; T2: immediately after Phase 1 intervention; T3: before Phase 2 intervention; T4: immediately after Phase 2 intervention, and completed the assessments within 1 week.
  Read records from nursing care daily record of the institutions.

CONTACTS AND LOCATIONS:
Overall Officials: Senyeong Kao, Ph.D, Study Chair — National Defense Medical Center, School of Public Health
Locations (1):
- Cardinal Tein Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liao CD, Lee PH, Hsiao DJ, Huang SW, Tsauo JY, Chen HC, Liou TH. Effects of Protein Supplementation Combined with Exercise Intervention on Frailty Indices, Body Composition, and Physical Function in Frail Older Adults. Nutrients. 2018 Dec 4;10(12):1916. doi: 10.3390/nu10121916. PMID 30518122
- [Result] Carlsson M, Littbrand H, Gustafson Y, Lundin-Olsson L, Lindelof N, Rosendahl E, Haglin L. Effects of high-intensity exercise and protein supplement on muscle mass in ADL dependent older people with and without malnutrition: a randomized controlled trial. J Nutr Health Aging. 2011 Aug;15(7):554-60. doi: 10.1007/s12603-011-0017-5. PMID 21808934